CLINICAL TRIAL: NCT00212108
Title: A Study Of Nasopharyngeal Carcinoma (NPC) Treated With Celecoxib And ZD1839
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Ross Soo, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP01/07/03
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: celecoxib, NPC, gefitinib
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Celecoxib; Gefitinib

ARMS (1):
- Celecoxib and ZD1839 (Experimental): Celecoxib and ZD1839 will be given twice a day and daily respectively for two consecutive weeks prior to further anti-cancer treatment.
  Interventions: Drug: celecoxib, gefitinib

INTERVENTIONS:
Drug: celecoxib, gefitinib — The dose of ZD1839 to be administered is 250mg. ZD1839 will be taken once daily in the morning at approximately the same time each day. If the patient inadvertently did not take the dose in the morning, the patient may take that dose anytime up to 10pm that same day. The daily treatment will be resumed the next day at the scheduled morning dose. Celecoxib will be administered at 400 mg bd.
  Other Names: ZD1839 (Iressa™)

SUMMARY:
EGFR and COX-2 are involved in tumorigenesis, angiogenesis and metastases and are frequently over expressed in NPC.COX-2 and EGFR inhibitors are active in NPC.There is synergistic action between COX-2 and EGFR inhibitors.

Study hypothesis: Celecoxib and gefitinib can reduce angiogenesis and induce anti-tumorigenicity in patients with nasopharngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven NPC.
2. Any clinical stage NPC as defined by the AJCC/UICC System.
3. No prior radiotherapy, chemoradiotherapy, immunotherapy or investigational agents.
4. No prior NSAIDs or corticosteroids for at least 4 weeks.
5. ECOG performance status ≤ 2.
6. Adequate end organ function
7. Life expectancy > 3 months.
8. Signed informed consent -

Exclusion Criteria:

1. Inability to take celecoxib and gefitinib for the specified period of time (14 days) prior to definitive therapy.
2. Tumor not visible on fibre nasopharyngoscopy for biopsy.
3. Known peptic ulcer disease.
4. Evidence of clinically active interstitial lung disease.
5. Previous or concomitant malignancies with the exception of adequately treated carcinoma-in-situ of the cervix and basal or squamous cell carcinoma of the skin.
6. Women who are pregnant or lactating. Females with child-bearing potential must have a negative serum pregnancy test within 7 days prior to study enrolment.
7. Women of childbearing potential who are not practising adequate contraception.
8. Concurrent medical problems that would significantly limit compliance with the study.
9. Presence of any underlying medical conditions (eg. Unstable or uncompensated respiratory, cardiac, renal or hepatic disease) that in the opinion of the investigator would make the patient unsuitable for study participation.
10. Known hypersensitivity to celecoxib and gefitinib or any of the excipients of the products, known sulphonamide sensitivity and allergic reaction following the ingestion of NSAIDs.
11. Known HIV, HBV or HCV infection. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-11; Primary Completion 2007-03 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To study histopathological changes in tumor following inhibition with celecoxib and gefitinib. | 1 year

SECONDARY OUTCOMES:
To evaluate the safety profile of celecoxib and ZD1839. | 30 days
To assess the pharmacokinetics of ZD1839 and celecoxib. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ross Soo, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore